CLINICAL TRIAL: NCT03315195
Title: A Randomized Controlled Trial Comparing Postoperative Complication Between Preoperative Oral Nutritional Supplement With Dietary Advice and Conventional Dietary Advice Alone in Patients Undergoing Elective Major Gastrointestinal Surgery
Brief Title: Preoperative Oral Nutritional Supplement vs Conventional Dietary Advice in Major Gastrointestinal Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Collaborators: Ramathibodi Hospital (Other)
Responsible Party: Principal Investigator, Narongsak Rungsakulkij, Lecturer, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ID 06-60-72
Record Dates: First submitted 2017-10-05; First posted 2017-10-20 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Surgery--Complications; Nutrition Aspect of Cancer
MeSH Terms: interventions — Dietary Supplements

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Preoperative oral nutritional supplement (Experimental): Oral nutritional supplement 500 kcal/day for 14 days and dietary advice
  Interventions: Dietary Supplement: Oral nutritional supplement (ONS)
- Conventional treatment (No Intervention): Dietary advice

INTERVENTIONS:
Dietary Supplement: Oral nutritional supplement (ONS) — ONS supplement by 500 kcal/day for 14 days
  Other Names: Nutren
  Arms: Preoperative oral nutritional supplement

SUMMARY:
Surgical outcome is associated the nutritional status of the patients. Perioperative nutritional supplement for malnutritional patient were recommended. There are several guidelines were recommended the perioperative nutrition for malnutrition patients. But in our hospital, there are no consensus guideline applied for the clinical practice. The nutritional supplement was judged by only attending physical This study was conducted to comparing the perioperative nutritional supplement with oral supplement with conventional approach with only dietary advice alone for all patients who undergoing major gastrointestinal surgery.

DETAILED DESCRIPTION:
The study design is a randomized controlled study. The eligible criteria is all patients who undergoing major gastrointestinal surgery including upper/lower gastrointestinal tract and hepatobiliary and pancratic surgery. After the informed consent are obtained. The patients are randomized into two group (study group and conventional group). The perioperative supplement with oral nutritional support and dietary advice were assigned in the study group. The conventional group were assigned only dietary advice. The blood test and nutritional assessment are performed by investigators in all participants. The participants were assessed two times before the operation (at first assigned and the day before the operation). The duration of nutritional supplement is at least fourteen days.The patient characteristic data, surgical intervention, and postoperative data were collected. The main outcome is the postoperative morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 year
* undergoing major gastrointestinal surgery
* able to take oral diet

Exclusion Criteria:

* unable to take oral diet
* Gastrointestinal tract insufficiency eg. gastrointestinal obstruction, perforation, malabsorption and peritonitis
* allergy to milk
* history of previous nutritional supplement from other source within one months
* chronic kidney disease (eGFR < 60 ml/min/1.73 m2)
* Take preoperative supplement less than 14 days
* Refused or withdraw from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 268 (Estimated)
Dates: Start 2017-11-25 (Actual); Primary Completion 2021-11 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Postoperative complications | 30 days after operation
  Number of complications

CONTACTS AND LOCATIONS:
Overall Officials: Narongsak Rungsakulkij, MD., Principal Investigator — Faculty of Medicine, Ramathibodi Hospital, Mahidol University, Thailand
Locations (1):
- Ramathibodi Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Komindrg S, Tangsermwong T, Janepanish P. Simplified malnutrition tool for Thai patients. Asia Pac J Clin Nutr. 2013;22(4):516-21. doi: 10.6133/apjcn.2013.22.4.06. PMID 24231010
- [Background] Antoun S, Rey A, Beal J, Montange F, Pressoir M, Vasson MP, Dupoiron D, Gourdiat-Borye A, Guillaume A, Maget B, Nitenberg G, Raynard B, Bachmann P. Nutritional risk factors in planned oncologic surgery: what clinical and biological parameters should be routinely used? World J Surg. 2009 Aug;33(8):1633-40. doi: 10.1007/s00268-009-0033-3. PMID 19387725
- [Result] Bozzetti F, Gianotti L, Braga M, Di Carlo V, Mariani L. Postoperative complications in gastrointestinal cancer patients: the joint role of the nutritional status and the nutritional support. Clin Nutr. 2007 Dec;26(6):698-709. doi: 10.1016/j.clnu.2007.06.009. Epub 2007 Aug 1. PMID 17683831
- [Result] Lohsiriwat V, Lohsiriwat D, Boonnuch W, Chinswangwatanakul V, Akaraviputh T, Lert-Akayamanee N. Pre-operative hypoalbuminemia is a major risk factor for postoperative complications following rectal cancer surgery. World J Gastroenterol. 2008 Feb 28;14(8):1248-51. doi: 10.3748/wjg.14.1248. PMID 18300352
- [Result] Szczepanik AM, Scislo L, Scully T, Walewska E, Siedlar M, Kolodziejczyk P, Lenart M, Rutkowska M, Galas A, Czupryna A, Kulig J. IL-6 serum levels predict postoperative morbidity in gastric cancer patients. Gastric Cancer. 2011 Aug;14(3):266-73. doi: 10.1007/s10120-011-0039-z. Epub 2011 Apr 20. PMID 21505767
- [Result] Argiles JM. Cancer-associated malnutrition. Eur J Oncol Nurs. 2005;9 Suppl 2:S39-50. doi: 10.1016/j.ejon.2005.09.006. PMID 16437757
- [Result] Garth AK, Newsome CM, Simmance N, Crowe TC. Nutritional status, nutrition practices and post-operative complications in patients with gastrointestinal cancer. J Hum Nutr Diet. 2010 Aug;23(4):393-401. doi: 10.1111/j.1365-277X.2010.01058.x. Epub 2010 Mar 23. PMID 20337847
- [Result] Kuzu MA, Terzioglu H, Genc V, Erkek AB, Ozban M, Sonyurek P, Elhan AH, Torun N. Preoperative nutritional risk assessment in predicting postoperative outcome in patients undergoing major surgery. World J Surg. 2006 Mar;30(3):378-90. doi: 10.1007/s00268-005-0163-1. PMID 16479353
- [Result] Baldwin C, Weekes CE. Dietary advice with or without oral nutritional supplements for disease-related malnutrition in adults. Cochrane Database Syst Rev. 2011 Sep 7;2011(9):CD002008. doi: 10.1002/14651858.CD002008.pub4. PMID 21901680
- [Result] Burden S, Todd C, Hill J, Lal S. Pre-operative nutrition support in patients undergoing gastrointestinal surgery. Cochrane Database Syst Rev. 2012 Nov 14;11:CD008879. doi: 10.1002/14651858.CD008879.pub2. PMID 23152265
- [Result] Kabata P, Jastrzebski T, Kakol M, Krol K, Bobowicz M, Kosowska A, Jaskiewicz J. Preoperative nutritional support in cancer patients with no clinical signs of malnutrition--prospective randomized controlled trial. Support Care Cancer. 2015 Feb;23(2):365-70. doi: 10.1007/s00520-014-2363-4. Epub 2014 Aug 6. PMID 25091056
- [Result] Parsons EL, Stratton RJ, Cawood AL, Smith TR, Elia M. Oral nutritional supplements in a randomised trial are more effective than dietary advice at improving quality of life in malnourished care home residents. Clin Nutr. 2017 Feb;36(1):134-142. doi: 10.1016/j.clnu.2016.01.002. Epub 2016 Jan 11. PMID 26847947
- [Result] Song GM, Tian X, Zhang L, Ou YX, Yi LJ, Shuai T, Zhou JG, Zeng Z, Yang HL. Immunonutrition Support for Patients Undergoing Surgery for Gastrointestinal Malignancy: Preoperative, Postoperative, or Perioperative? A Bayesian Network Meta-Analysis of Randomized Controlled Trials. Medicine (Baltimore). 2015 Jul;94(29):e1225. doi: 10.1097/MD.0000000000001225. PMID 26200648
- [Result] Burden ST, Gibson DJ, Lal S, Hill J, Pilling M, Soop M, Ramesh A, Todd C. Pre-operative oral nutritional supplementation with dietary advice versus dietary advice alone in weight-losing patients with colorectal cancer: single-blind randomized controlled trial. J Cachexia Sarcopenia Muscle. 2017 Jun;8(3):437-446. doi: 10.1002/jcsm.12170. Epub 2017 Jan 3. PMID 28052576
- [Result] Kondrup J, Allison SP, Elia M, Vellas B, Plauth M; Educational and Clinical Practice Committee, European Society of Parenteral and Enteral Nutrition (ESPEN). ESPEN guidelines for nutrition screening 2002. Clin Nutr. 2003 Aug;22(4):415-21. doi: 10.1016/s0261-5614(03)00098-0. PMID 12880610
- [Result] Kondrup J, Rasmussen HH, Hamberg O, Stanga Z; Ad Hoc ESPEN Working Group. Nutritional risk screening (NRS 2002): a new method based on an analysis of controlled clinical trials. Clin Nutr. 2003 Jun;22(3):321-36. doi: 10.1016/s0261-5614(02)00214-5. PMID 12765673
- [Result] Weimann A, Braga M, Harsanyi L, Laviano A, Ljungqvist O, Soeters P; DGEM (German Society for Nutritional Medicine); Jauch KW, Kemen M, Hiesmayr JM, Horbach T, Kuse ER, Vestweber KH; ESPEN (European Society for Parenteral and Enteral Nutrition). ESPEN Guidelines on Enteral Nutrition: Surgery including organ transplantation. Clin Nutr. 2006 Apr;25(2):224-44. doi: 10.1016/j.clnu.2006.01.015. Epub 2006 May 15. PMID 16698152